CLINICAL TRIAL: NCT01204827
Title: Follow Up of Patients With HBeAg Negative Chronic Hepatitis B Virus Infection Treated With Sebivo (Telbivudine) Using the 13C Methacetin Breath Test (BreathID®)
Brief Title: Follow Up of Patients Chronic Hepatitis B (CHB) Treated With Sebivo Using the 13C Methacetin Breath Test
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Hadassah Medical Organiztion, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: CLDT600AIL02T
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Hepatitis B
Keywords: Patients with chronic HBeAg negative hepatitis B virus infection treated with Sebivo (Telbivudine)
MeSH Terms: conditions — Hepatitis B, Chronic

ARMS (1):
- CHBV Sebivo (Experimental)
  Interventions: Device: 13C Methacetin Breath Test (BreathID)

INTERVENTIONS:
Device: 13C Methacetin Breath Test (BreathID)

SUMMARY:
Patients with HBeAg negative chronic HBV and evidence of hepatic disease (elevated liver enzymes or evidence of cirrhosis) who have significant viremia are treated with anti HBV therapy. Currently the key goals of anti HBV therapy are profound and prolonged viral suppression and treatment efficacy is assessed by monitoring viral load and liver enzymes. However these do not always reflect the degree of liver impairment or the degree of improvement in response to therapy. Sebivo has been accepted in Israel as a first line therapy for HBeAg negative and HBeAg positive chronic HBV with evidence of liver damage. Viral load should decrease by 1 log every 3 months, otherwise patients should be offered add-on or alternative therapy. As the majority of patients in Israel are HBeAg negative chronic HBV and in order to have homogenous population we will select for our study only patients with HBeAg negative chronic HBV. The 13C Methacetin breath test, assess liver function and specifically the function of the microsomal CYP4501A2. It has been shown to correlate with the degree of liver impairment and with clinical outcomes in both acute and chronic liver disease. The aim of this study is to determine the utility of the 13C Methacetin Breath Test to follow up patients with HBeAg negative chronic HBV receiving anti viral therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age.
2. Documented chronic hepatitis B (CHB) infection defined by all of the following:

   * Clinical history compatible with CHB
   * HBeAg negative chronic hepatitis B patients
   * Detectable serum HBsAg at least 6 months prior to screening
   * Serum HBV DNA level ≥ 2000 IU/mL as determined by either the Abbott or Roche Taqman assay at Screening visit
   * For patients with cirrhosis, clinical history and lab tests compatible with compensated liver disease
   * Elevated serum ALT level > x 1 ULN and < x 10 ULN) at Screening visit (ULN being 30 IU/mL)
   * If ALT level ≤ x 1 ULN must have available liver histology report within 12 months before screening which indicates chronic hepatitis. If not available, liver biopsy is required at baseline.
3. Patient is willing and able to comply with the study drug regimen and all other study requirements.
4. The patient is willing and able to provide written informed consent to participate in the study.

Exclusion Criteria:

1. History of hypersensitivity to any of the study drugs (Methacetin, Sebivo) or to drugs with similar chemical structures, including allergy to paracetamol.
2. Patient is pregnant or breastfeeding.
3. Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means. The exception of the aforementioned criteria will be given if they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/ml (IU/L) or 6 weeks post surgical bilateral oophorectomy with or without hysterectomy or have been surgically sterilized (e.g., bilateral tubal ligation) or the patient must agree to use two methods of birth control. This is any combination of hormonal contraception (implantable, patch, oral or injection), IUD, male or female condom with spermicidal gel, diaphragm, sponge or cervical cap. Women of childbearing potential must have a negative serum betahuman chorionic gonadotropin (β-HCG) during
4. Males capable of reproduction, defined as all men physiologically capable of producing sperm, including men whose career, lifestyle, or sexual orientation precludes intercourse with a female partner UNLESS the female partner meets the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/ml (IU/L) or the patient must agree to use two methods of birth control. This is any combination of hormonal contraception (implantable, patch ,oral or injection), IUD, male or female condom with spermicidal gel, diaphragm, sponge or cervical cap.
5. Patient is co-infected with HCV, HDV, or HIV.
6. Severe uncontrolled disease of other organ (heart, kidney, lung).
7. Patients who have previously been involved in a trial with telbivudine.
8. Patient has received nucleoside or nucleotide drugs whether approved or investigational at any time.
9. Patient has received IFN or other immunomodulatory treatment in the 6 months before Screening for this study.
10. Patient has a history of or clinical signs/symptoms of hepatic decompensation such as ascites, esophageal variceal bleeding, hepatic encephalopathy, hepatorenal syndrome, hepatic hydrothorax, hepatopulmonary syndrome or spontaneous bacterial peritonitis, among others.
11. Patient has a medical condition that requires prolonged or frequent use of systemic acyclovir or famciclovir.
12. Patient has a history of malignancy of any organ system, treated or untreated, within the past 5 years whether or evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin. Patients with previous findings suggestive of possible hepatocellular carcinoma (HCC), should have the disease ruled out prior to entrance into the study.
13. Patient has one or more additional known primary or secondary causes of liver disease other than CHB, including steatohepatitis and autoimmune hepatitis among other liver diseases. Gilbert's syndrome and Dubin-Johnson syndrome are not considered exclusion criteria for this study.
14. History of any other acute or chronic medical condition that in the opinion of the investigator would make the patient unsuitable for inclusion into the study.
15. Patient is currently abusing alcohol or illicit drugs, or has a history of alcohol abuse or illicit substance abuse within the preceding two years.
16. Patient has a medical condition that requires frequent or prolonged use of systemic corticosteroids, although inhaled corticosteroids are allowed.
17. Patient has a history of clinical and laboratory evidence of chronic renal insufficiency (Estimated calculated serum creatinine clearance < 50)
18. Patient has a medical condition requiring the chronic or prolonged use of potentially hepatotoxic drugs or nephrotoxic drugs.
19. Patient has any other concurrent medical or social condition likely to preclude compliance with the schedule of evaluations in the protocol, or likely to confound the efficacy or safety observations of the study.
20. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
21. Patient has a history of myopathy, myositis, or persistent muscle weakness.
22. Patient has any of the following laboratory values during Screening:

    * Hemoglobin <11 g/dL (110 g/L) for men or <10 g/dL (100 g/L) for women
    * Total WBC <3,500/mm3 (3.5 x 109/Liter)
    * Absolute neutrophil count (ANC) <1,500/mm3 (1.5 x 109/Liter)
    * Platelet count <75,000/mm3 (75 x 109/Liter)
    * Serum amylases or lipase ≥ 1.5 x ULN
    * Serum albumin <3.3 g/dL (33g/L)
    * Total bilirubin ≥ 2.0 mg/dL (34.2 μmol/L)
    * Estimated calculated serum creatinine clearance < 50 mL/min ( 0.48 ml/s) using the Cockcroft-Gault method with lean or ideal body weight; see Glossary of Terms (Cockcroft 1976)
    * AFP > 50 ng/mL or μg/L (requires further work up per local medical standards)
23. Patient has not fasted for 8 hours.
24. Patient has smoked on the day of the test.
25. Patient that has taken drugs that can interfere with methacetin metabolism: fluvoxamine, amiodarone, ciprofloxacin, cimetidine, rifampin, carbamazepine within the last 24 hours.
26. Patient has taken Tylenol or any other acetaminophen related medications within the past 24 hours.
27. Patients that received any new medication in the last 48 hours.
28. Patients that still suffer from any previous clinical intervention (e.g. biopsy)
29. Patients who have not consumed alcohol 24 hours prior the MBT or consume alcohol on a regular basis more than 40gr for male and 20gr for female per day.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Unit, Hadassah Hebrew University Medical Center, Jerusalem, Israel